CLINICAL TRIAL: NCT01492608
Title: Administration of Antenatal Magnesium Sulphate for Prevention of Cerebral Palsy and Death in Preterm Infants (MASP-STUDY)
Brief Title: Magnesium Sulphate for Preterm Birth (MASP Study)
Acronym: MASP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Lene Huusom, Medical Doctor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT number 2011-000735-80; Projectnumber 2010-382 (Registry Identifier: The Danish Committee on Biomedical Research Ethics)
Record Dates: First submitted 2011-12-11; First posted 2011-12-15 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
Keywords: magnesium sulphate; preterm birth; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Premature Birth | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulphate (Active Comparator): Magnesium sulphate will be given as a loading dose of 5 g infused for 20-30 minutes, followed by a maintenance dose of 1 g per hour. Placebo will be given in identical appearing doses. The maintenance infusion will be continued until delivery appears, or for 24 hours if delivery does not occur or no longer is considered imminent. The infusion will be resumed when delivery is considered imminent again. Another loading dose of 5 g will be given if at least 6 hours has passed after infusion was stopped. The doses that are used in this project are similar to those used for prevention of eclampsia among women with severe preeclampsia.
  Interventions: Drug: Magnesium sulphate
- Natriumchlorid (Placebo Comparator): Placebo and the active drug (Magnesium sulphate) will be administered identically (same loading and maintenance dose for the same period of time).
  Interventions: Drug: Magnesium sulphate

INTERVENTIONS:
Drug: Magnesium sulphate — Magnesium sulphate will be given as a loading dose of 5 g infused for 20-30 minutes, followed by a maintenance dose of 1 g per hour. Placebo will be given in identical appearing doses. The maintenance infusion will be continued until delivery appears, or for 24 hours if delivery does not occur or no longer is considered imminent. The infusion will be resumed when delivery is considered imminent again. Another loading dose of 5 g will be given if at least 6 hours has passed after infusion was stopped. The doses that are used in this project are similar to those used for prevention of eclampsia among women with severe preeclampsia.
  Other Names: Magnesium sulfat

SUMMARY:
The purpose of the study is to assess whether magnesium sulphate for women at risk of preterm birth can protect their children against cerebral palsy. The results from this randomised controlled trial will be added to the previous meta-analysis to obtain firm evidence for magnesium sulphate as a neuroprotector, and determine whether it should be used as standard therapy for women in preterm birth.

DETAILED DESCRIPTION:
Cerebral palsy consists of chronic and non-progressive clinical syndromes that are characterized by motor and postural dysfunction. In affected infants, voluntary movements become difficult and limited, and although clinical expression may change with time, this disability is accompanied with major personal and socioeconomic burdens. Preterm infants have increased risk of cerebral palsy, which is inversely correlated with gestational age at birth.

Previous studies have indicated that magnesium sulphate may be neuroprotective for the preterm infant, when the drug is given to women prior to preterm birth.

However, this benefit of antenatal magnesium sulphate was recently questioned by Trial Sequential Analysis (TSA), a statistical method that adjusts for risk of random error on published meta-analyses. TSA demonstrates that additional data are needed before accepting magnesium sulphate as evidence based therapy for women in preterm labour. Therefore we will close the gap by performing a new randomised clinical trial (RCT), which aims to assess whether magnesium sulphate for women prior to preterm birth can protect their children against cerebral palsy.

The RCT will not individually have the power to detect a significant difference between magnesium and placebo. Instead, when the trial is completed, the results will be added to the previous meta-analysis to obtain firm evidence for magnesium sulphate as a neuroprotector, and determine whether it should be used as standard therapy for women in preterm birth.

From Denmark 560 eligible women, who are at risk of preterm birth at 24 to 32 weeks of gestation, will be randomised to receive either intravenous magnesium sulphate or placebo. Randomisation will be performed blinded by computer generated random numbers.

The children are followed up by medical records and by Ages and Stages Questionnaire (ASQ) in the age of 18 month or older. To screen for cerebral palsy, the domains gross motor skills and fine motor skills are together with the total score the most suitable measures.

1. If the medical record is without any information on cerebral palsy and/or delayed motor development or if there is no medical record to be found and there is an ASQ score above the 20% percentile (in the domains of gross motor function, fine motor function or total score), the child is classified as not having cerebral palsy.
2. If the child in the ASQ scores under the 20% percentile in the domains of gross motor function, fine motor function and/or total score and there is no diagnosis of cerebral palsy in the medical record, the parents are contacted. The parents are contacted as well, if there is no medical record to be found. If the parents explain that the child is developing normally and is not seen by doctors or physiotherapists, the child is classified as not having cerebral palsy. If the parents state that the child is not developing normally, the child is invited to further examination by a pediatric neurologist.
3. If the child is diagnosed with cerebral palsy or delayed motor development, the medical journal is reviewed by a pediatric neurologist to verify the diagnosis. If there is any doubt about the correctness of the diagnosis, the child is invited to further examination by a pediatric neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24+0-31+6 weeks
* Singletons or twins
* Preterm rupture of membranes at 24+0-31+6 weeks with contractions and expected birth within 2-24 hours
* Preterm contractions and expected birth within 2-24 hours
* Anticipated delivery within 2-24 hours of other reasons (due to for example fetal growth restriction)
* Age 18 years at inclusion

Exclusion Criteria:

* Major fetal abnormalities or fetal death. (Major fetal abnormalities are chromosome abnormalities, myelomeningocele and cerebral abnormalities that gives neurological handicaps)
* Maternal contraindication to magnesium sulphate (for example pulmonary disorders, kidney diseases with creatinin > 100, myasthenia gravis, atrioventricular block, treatment with aminoglycosides)
* Magnesium sulphate given for other reasons (for example for prevention of eclampsia)
* Patients who do not speak and understand Danish
* Allergies towards magnesium sulphate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 560 (Actual)
Dates: Start 2011-12-16 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Moderate or severe cerebral palsy | At 18 months of age
  The difference in the number of children with moderate or severe cerebral palsy at 18 months of age, whose mothers had magnesium sulphate before birth compared to the group of children whose mothers received placebo before birth.

SECONDARY OUTCOMES:
Perinatal death | From date of randomization until the date of death from any cause, assessed up to 18 months
  The difference in the number of children with perinatal death, whose mothers had magnesium sulphate before birth compared to the group of children whose mothers received placebo before birth.
Composite outcome of outcome 1 and 2 (moderate-severe cerebral palsy and perinatal death) | At 18 months of age
  Frequency of the composite outcome in the two groups ((intervention and placebo group)
Blindness | At 18 months of age
  The difference in the number of children with blindness at 18 months of age, whose mothers had magnesium sulphate before birth compared to the group of children whose mothers received placebo before birth.
Apgar scores | At 1 minute and 5 minutes after birth
  The difference in apgar scores in the group of children, whose mothers had magnesium sulphate before birth compared to the group of children whose mothers received placebo before birth.

OTHER OUTCOMES:
Cranial ultrasound findings | Assessed up to 18 months of age
  Frequency of intraventricular hemorrhage and periventricular leukomalacia in the two groups ((intervention and placebo group).
Resuscitation in delivery room | First hour of life
  Mode of resuscitation in delivery room in the two groups (intervention and placebo group)
Neonatal convulsions | Assessed up to 18 months of age
  Clinically verified convulsions during first neonatal admission.
Use of respiratory support | Assessed up to 18 months of age
  Endotracheal ventilation or continuous positive airways pressure, or both during first neonatal admission.
Bronchopulmonary dysplasia (BPD) | Assessed up to 18 months of age
  Mild BPD: Need for continuous, supplemental oxygen at ≥ 28 days but not at 36-week postmenstrual age.
  Moderate BPD: Need for continuous, supplemental oxygen at 28 days, in addition to supplemental oxygen at ≤30% at 36-week postmenstrual age.
  Severe BPD: Need for continuous, supplemental oxygen at 28 days and, at 36-week postmenstrual age, the need for mechanical ventilation and/or oxygen >30%
Hypotension | Assessed up to 18 months of age
  Need of volume therapy or vasopressors during first neonatal admission.
Length of neonatal hospitalization | Assessed up to 18 months of age
  Length of the neonatal hospitalization measured in days. From time of birth to discharge after first neonatal admisson or until death.
Retinopathy of prematurity | At 18 months of age
  Retinopathy of prematurity stage 1-5
Patent ductus arteriosus | At 18 months of age
  Ultrasound verified patent ductus arteriosus
Necrotizing enterocolitis | Assessed up to 18 months of age
  Defined according to Bell's critiria
Cerebral palsy | At 18 months of age
  Mild (GMFCS level I), moderate (II-III), severe (IV-V), any
Blood transfusion | Assessed up to 18 months of age
  Number of children receiving bood transfusion during first admission
Deafness | At 18 months of age
  One or both ears

CONTACTS AND LOCATIONS:
Overall Officials: Lene Huusom, MD, Principal Investigator — Department of Gynecology and Obstetrics, Hvidovre Hospital, Denmark
Locations (14):
- Denmark (14):
  - Hanne Trap Wolf, Hvidovre, Danmark
  - Gynækologisk afdeling D, Odense, Fyn
  - Gynækologisk-Obstetrisk Afdeling, Aalborg, Jylland
  - Gynækologisk-obstetrisk afdeling Y, Aarhus, Jylland
  - Gynækologisk obstetrisk Afdeling, Esbjerg, Jylland
  - Gynækologisk-obstetrisk afd., Kolding, Jylland
  - Gynækologisk obstetrisk afdeling, Randers, Jylland
  - Gynækologisk-obstetrisk afd., Silkeborg, Jylland
  - Kvindeafdeling Y, Viborg, Jylland
  - Obstetrisk Klinik, Copenhagen, Region Sjælland
  - Gynækologisk Obstetrisk afdeling, Herlev, Region Sjælland
  - Gynækologisk-Obstetrisk Afdeling, Hillerød, Region Sjælland
  - Gynækologisk Obstetrisk afdeling, Holbæk, Region Sjælland
  - Gynækologisk-obstetrisk afdeling, Næstved, Region Sjælland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huusom LD, Secher NJ, Pryds O, Whitfield K, Gluud C, Brok J. Antenatal magnesium sulphate may prevent cerebral palsy in preterm infants--but are we convinced? Evaluation of an apparently conclusive meta-analysis with trial sequential analysis. BJOG. 2011 Jan;118(1):1-5. doi: 10.1111/j.1471-0528.2010.02782.x. No abstract available. PMID 21197681

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT01492608/SAP_000.pdf